CLINICAL TRIAL: NCT05762484
Title: The Efficacy of Laser Hair Removal Therapy in Patients With Mild to Moderate HS, a Randomized Controlled Trial.
Brief Title: Efficacy of Laser Hair Removal Therapy in HS
Acronym: HaLa
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Hessel H van der Zee, MD, PhD, MD, PhD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMCD_22026
Record Dates: First submitted 2022-12-23; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Hidradenitis Suppurativa, Acne Inversa
Keywords: laser hair removal therapy
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Clindamycin

STUDY DESIGN:
Intervention Model Description: RCT with intervention and control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group, laser hair removal therapy (Experimental): Patients will undergo 6 monthly laser hair removal treatments with de Nd:YAG laser. After 6 months, a 6 follow up will start, using clindamycin 1% lotion if needed.
  Interventions: Procedure: Nd:YAG laser hair removal
- Control group, clindamycin 1% lotion if needed, standard care (Active Comparator): Patients will use clindamycin 1% lotion of needed for 1 year.
  Interventions: Drug: Clindamycin 1 % Topical Lotion

INTERVENTIONS:
Procedure: Nd:YAG laser hair removal — Using the Nd:YAG laser (cynergy), hair of the axillae will be removed.
  Arms: Intervention group, laser hair removal therapy
Drug: Clindamycin 1 % Topical Lotion — Clindamycin 1% lotion if needed
  Arms: Control group, clindamycin 1% lotion if needed, standard care

SUMMARY:
Hidradenitis suppurativa (HS) is a chronic, recurrent and debilitating inflammatory skin disorder, characterized by painful inflamed nodules, abscesses and tunnels in the skin folds such as the axilla, inguinal region and gluteal area. The primary event in HS is occlusion of the hair follicle. HS is a notoriously difficult to treat disease, because treatment options are limited and evidence based treatments are scarce. Prevention of diseases is an important topic in medicine. However, current clinical trials in HS are focusing on anti-inflammatory drugs in patients with severe HS, whereas prevention and treatment of patients with more common mild HS is neglected. Laser hair removal therapy is a non-invasive procedure with minimal treatment discomfort for patients. Previous limited studies have suggested positive results in favor of laser hair removal therapy in HS. We therefore hypothesize that hair depilation using laser hair removal therapy may prevent the formation of new lesions and flares of the disease. The objective is to assess the efficacy of laser hair removal therapy in patients with mild to moderate HS.

ELIGIBILITY:
Inclusion Criteria:

* IHS4 mild to moderate, without tunnels in the axillae.
* HS activity in at least one axilla.
* Age 18 years and over.

Exclusion Criteria:

* If the patient is not able or willing to provide informed consent.
* If the patient is allergic to clindamycin lotion.
* If the patient uses systemic therapy for HS such as antibiotics or biologicals.
* If a patient is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Difference in IHS4 over time, measured between month 7 to month 12 | between month 7 to 12
  The IHS4 will be assessed monthly.

SECONDARY OUTCOMES:
Cumulative IHS4 over month 7 to month 12 between the two groups | month 7 to 12
  IHS4 will be calculated on a monthly bases. IHS4 will be added up per visit which makes it a cumulative outcome
Change in skin related pain of the axillae, on a numerical rating scale (NRS), between baseline and month 12, and between groups. | every month for 12 months
  NRS pain will be assessed
Change in skin related itch of the axillae, on a NRS, between baseline and month 12, and between groups. | every month for 12 months
  NRS itch will be assessed
Difference in number of self-reported flares (number of flares reported by the patients in the last 4 weeks), between the two groups during this study | every month for 12
  Number of self reported flares will be assessed
Difference and change in quality of life measured with the Dermatologic Life Quality Index (DLQI) between baseline and month 12 and between groups. | every month for 12 months
  PROM will be assessed
Difference and change in quality of life measured with the Hidradenitis Suppurativa Quality of Life score (HiSQOL), between baseline and month 12 and between groups. | every month for 12 months
  PROM will be assessed
Difference in patients satisfaction score at month 12 between groups. | every month for 12 months
  patients satisfaction will be assessed
Cumulative IHS4 over month 7 to 12, correlated to hair loss after six months. | every month for 12 months
  the amount of hair loss will be assessed and correlated to the cumulative IHS4
Cumulative IHS4 calculated over a time period of 3, 9 and 12 months between groups. | every month for 12 months
  The cumulative IHS4 will be assessed after 3, 9 and 12 months
Difference in pustule and papule count during visits over month 1 to 12 between groups. | every month for 12 months
  the number of papules and pustules will be assessed
Difference in (cumulative) abscess en nodule count over month 1 to 12 between groups. | every month for 12 months
  number of abscesses and nodules will be assessed
Difference in number of times escape medication has been used over month 1 to 12 between groups. | every month for 12months
  Number of escape medication will be assessed
Difference of average duration of a flare, reported by the patient, over month 1 to 12 between groups. | every month for 12 months
  Duration of a flare will be assessed
The difference in IHS4 and HS-PGA, measured every visit. | every month for 12 months
  The IHS4 and HS-PGA will be assessed
Amount of clindamycin lotion use for both groups. | every month for 12 months
  clindamycin 1% lotion will be weighted every visit
Difference in number of adverse events between groups. | every month for 12 months
  safety will be assessed using adverse events
Incidence and severity of all adverse events (according to medDRA) will be analysed throughout the study. | every month for 12 months
  safety will be assessed using adverse events
Histopathological: diameter hair shaft in axillary skin before and after treatment. | Measured at baseline (month 1), after laser hair removal therapy (month 7) and six months after laser hair removal therapy (month 12), for the intervention group
  Biopsies will be taken for histopathological research
Histopathological: plugging of the hair follicle in the skin before and after treatment | Measured at baseline (month 1), after laser hair removal therapy (month 7) and six months after laser hair removal therapy (month 12), for the intervention group
  Biopsies will be taken for histopathological research
Histopathological: immunohistochemistry in the skin before and after treatment | Measured at baseline (month 1), after laser hair removal therapy (month 7) and six months after laser hair removal therapy (month 12), for the intervention group
  Biopsies will be taken for histopathological research
Histopathological: AMP expression in the skin before and after treatment | Measured at baseline (month 1), after laser hair removal therapy (month 7) and six months after laser hair removal therapy (month 12), for the intervention group
  Biopsies will be taken for histopathological research

CONTACTS AND LOCATIONS:
Overall Officials: Hessel van der Zee, MD, PhD, Principal Investigator — Erasmus Medical Center

IPD SHARING:
Plan to Share IPD: Undecided